CLINICAL TRIAL: NCT05015075
Title: Role of Early Short-term Cardiac Rehabilitation in Patients Undergoing Pacemaker Implantation
Brief Title: Cardiac Rehabilitation After Pacemaker Implantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Principal Investigator, Jinhee Ahn, MD, Clinical associate professor, Pusan National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-1803-017-064
Record Dates: First submitted 2021-07-27; First posted 2021-08-20 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Bradycardia; Pacemaker
MeSH Terms: conditions — Bradycardia | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CR group (Experimental): participants who have exercise-based cardiac rehabilitation program after PM.
  Interventions: Behavioral: cardiac rehabilitation
- non-CR group (Placebo Comparator): participants who have only routine regular follow-up after PM instead of CR program
  Interventions: Behavioral: cardiac rehabilitation

INTERVENTIONS:
Behavioral: cardiac rehabilitation — cardiac rehabilitation after pacemaker implantation
  Other Names: exercise-based cardiac rehabilitation: step-box, lower extremity recumbent ergometer

SUMMARY:
The investigators assessed whether short-term cardiac rehabilitation following pacemaker implantation was enough to improve both physical function and quality of life.

DETAILED DESCRIPTION:
Exercise-based cardiac rehabilitation (CR) improves clinical outcomes in patients with cardiovascular diseases. However, few data exist regarding the role of early short-term CR in patients undergoing pacemaker (PM) implantation. The investigators assessed whether short-term CR following PM implantation was enough to improve both physical function and quality of life (QOL).

ELIGIBILITY:
Inclusion Criteria:

* patients who were scheduled to undergo new PM implantation

Exclusion Criteria:

* patients older than 75 years
* patients who are contraindicated to exercise
* patients who refuse to participate

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2019-01-11 (Actual); Study Completion 2019-08-17 (Actual)

PRIMARY OUTCOMES:
changes in physical function based on cardiopulmonary exercise test | 1 month
  VO2 max in mL/kg/min

SECONDARY OUTCOMES:
changes in physical function based on muscle power test | 1 month
  knee extension in kilogram
changes in quality of life | 1 month
  SF-36 questionnaire score

CONTACTS AND LOCATIONS:
Locations (1):
- Jinhee Ahn, Busan, South Korea